CLINICAL TRIAL: NCT04776174
Title: Crossover Comparison of the Efficacy and Tolerance of Telerobotic vs Standard Ultrasound Exam in Children
Brief Title: Efficacy and Tolerance of Telerobotic vs Standard Ultrasound Exam in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: ADECHOTECH (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHILDMELODY
Record Dates: First submitted 2021-02-08; First posted 2021-03-01 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Children will be initially scanned with a telerobotic ultrasound system. Within 3 hours after the telerobotic examination, patients will be scanned by a different sonographer with similar experience and qualifications using the conventional ultrasound, who will be blinded to the findings of the telerobotic examination.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- standard and telerobotic ultrasound (Experimental): Included patients will have both ultrasound examination: standard ultraosound (abdominal, cardiac or pulmonary depending on the prescription and telerobotic ultrasound
  Interventions: Device: Ultrasound using the telerobotic Melody system

INTERVENTIONS:
Device: Ultrasound using the telerobotic Melody system — The children will first have a telerobotic ultrasound abdominal, pulmonary or cardiac followed by a classical ultrasound.

SUMMARY:
In children with Covid-19, the diagnosis of Kawasaki Disease (KD) and pneumonia should be made very quickly. However, the regional hospitals surrounding Paris don't have the required expertise. The use of MELODY allows the paediatric team to quickly carry out the necessary examinations while avoiding the movement of patients and the risk of contamination.

The MELODY remote system developed by the company AdEchoTech is a CE marking telemedicine technique, allowing an expert to perform an ultrasound scan on a distant patient (several hundred/thousands of kms). The Melody system makes it possible to optimize ultrasound expertise resources wherever they are located (all specialties combined) The feasibility of the clinical use of telerobotic sonography has been demonstrated in adults for abdominal, cardiac and prenatal exam. Thus, the aim of this study is to assess the feasibility of this system in children.

ELIGIBILITY:
Inclusion Criteria:

* Patient from 1 year to 10 years
* Patient requiring an ultrasound exam (thoracic, abdominal or cardiac)
* French social security affiliation

Exclusion Criteria:

* Obesity defined by a BMI greater than 30
* Open wound making it impossible to carry out an ultrasound scan
* Algetic patient
* Instability of vital functions
* Impossible to remain in a seated position
* Refusal to participate in the study

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
Number of normal and abnormal standard and telerobotic ultrasound examinations | 1 day
  Number of normal and abnormal examination conclusion for telerobotic and conventional ultrasound examinations

SECONDARY OUTCOMES:
Age of participants | At baseline
  Age of patients with telerobotic ultrasound
Number of anomalies found | Up to 4 hours
  Conventional and telerobotic ultrasound examinations results
Parent satisfaction | Up to 4 hours
  Parent satisfaction questioner for the telerobotic examination using a 5-point Liekert scale from 1: "strongly disagree" to 5: "strongly agree"
Medical assistant satisfaction | Up to 4 hours
  Medical assistant satisfaction questioner for the telerobotic examination using a 5-point Liekert scale from 1: "strongly disagree" to 5: "strongly agree"
Sonographer satisfaction | Up to 4 hours
  Sonographer satisfaction questioner for the telerobotic examination using a 5-point Liekert scale from 1: "strongly disagree" to 5: "strongly agree"

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHI Créteil, Créteil
  - CHI Villeneuve-Saint-Georges, Villeneuve-Saint-Georges

IPD SHARING:
Plan to Share IPD: No